CLINICAL TRIAL: NCT04144452
Title: Effects of Therapeutic Exercises and Educational Sessions After Microdiscectomy Through Minimally Invasive Surgery for Disc Herniation
Brief Title: Therapeutic Exercises and Educational Sessions After Microdiscectomy for Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ghurki Trust and Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Minimally Invasive Surgical Procedures; Disk, Herniated
Keywords: Back Pain; Exercise Therapy; Functionality; Microdiscectomy; Patient Education; Quality of Life
MeSH Terms: conditions — Intervertebral Disc Displacement; Back Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Education Session (Active Comparator): Educational session will be given twice a day for three months. Individualized instructional booklet about back care for each patient will be designed, reviewed and finalized by operating surgeons according to the needs of patients.
  Interventions: Other: Patient Education Session
- Therapeutic exercises plus educational sessions (Experimental): Trunk and lower musculature strength and endurance training will be performed twice a week for three months. Therapeutic exercises incorporating mat exercises will be performed. Progression will be made according to patient status.
  Interventions: Other: Therapeutic Exercise plus educational session

INTERVENTIONS:
Other: Patient Education Session — The intervention of Patient Education will be designed individually according to the patient's need who have undergone lumbar microdiscectomy procedure through MIS. The basic purpose of the educational session will be to inform the participants about their pre operative and current back condition and discuss methods to care for their back. The session will be given for one hour and face to face interaction will be ensured twice a week. Initially the post operative education plan and instructions will be formulated, reviewed and finalized by the operating surgeon.
  Arms: Patient Education Session
Other: Therapeutic Exercise plus educational session — Therapeutic exercises include strength and endurance training and mat exercises. Strengthening exercises of the trunk extensors will be initiated first and then endurance exercises will be targeted. Mat exercises will be performed to strengthen the back and lower musculature. Treatment will be given twice a week for almost three months. Individualized educational sessions will be performed in the same way as conducted in the other group. Progression of the exercises and the rest periods will be incorporated according to the status of patient.
  Arms: Therapeutic exercises plus educational sessions

SUMMARY:
The basic purpose of current research is to evaluate the comparative effectiveness of therapeutic exercises and educational sessions after microdiscectomy through Minimally Invasive Surgery for disc herniation. A Randomized trial will be conducted on 60 patients from Ghurki hospital , divided into two groups. Simple random sampling will be utilized as sampling strategy. Assessment of physical activities of daily living and quality of life will be performed before and after 8 weeks of post intervention surgery through Oswestry Disability Index, Physical activity survey , SF 36 and Subjective Quality of Life scale respectively . A follow up assessment will be performed after 6 months. Analysis will be done through SPSS 21.

DETAILED DESCRIPTION:
The increasing number of spinal injuries and pathologies directs the need of technological advancement in spinal surgeries and its approaches in Pakistan. Among various expansion in surgical procedures; minimally invasive surgery of spine has gaining more advantage for spinal decompression, spinal fusion and instrumentation over lumbar, thoracic and cervical spine areas considering multilevel pathology.(1) Minimally invasive spine surgery (MISS), has attracted increasing attention within the last decade. The common thread between all minimally invasive spine surgeries is use of smaller incisions and less deterioration of surrounding soft tissue, typically results in less pain after surgery and a faster recovery with reduced length of stay at hospital. The patient reported functional outcome after this procedure was found to be better in comparison with the open approach procedures.(2) Therapeutic exercise post-operatively was programmed to maximize recovery and to minimize potential future problems including disability and improving quality of life. Three different approaches for post-operative management has been practiced including: 1. Recovery phase: 4 to 16 weeks of limited activity following the surgery, 2. eliminating post-operative activity restriction leads to enhanced short-term outcomes for patients after limited open discectomy, 3. Incorporating therapeutic exercise intervention program.(3) The purpose of therapeutic exercise post-operatively was to maximize recovery and to minimize potential future problems including disability and improving quality of life. (4)The therapeutic intervention program comprises of two components: patient education and exercise therapy based on protocols by clinical expertise considering the philosophy of surgeon. Patient education comprises of a one hour counseling session. Therapeutic exercise program encompasses trunk strengthening exercises (both isometrics and dynamics) along with core stabilization exercises and endurance training. (5)

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 to 50 years
* Diagnosed cases of L4-L5 through Gold standard MRI
* Who have undergone minimally invasive microdiscectomy due to herniated disc
* Both male and female
* Patients who will be without adverse events or complications 4 weeks post surgery

Exclusion Criteria:

* Low back pain due to causes other than herniated disc
* Leg pain due to causes other than herniated disc
* Who have undergone standard/open microdiscectomy
* Previous history of spinal surgery
* Patients unwilling to participate

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Post Surgery (Oswestry Disability Questionnaire) | 3 months
  The Oswestry Disability Index is considered as a vital tool that investigators and disability assessors use to measure an individual's permanent functional disability. The test is defined as the 'gold standard' of low back functional outcome tools.
  ODI consist of 10 items and each item is scored on Likert scale from 0 to 5. The total score is then added and multiplied by 2. Thus the score is from 0 to 100. Greater score represents more severe disability.

SECONDARY OUTCOMES:
Change from Baseline Post Surgery (Short Form 36) | 3 months
  Short Form -36 will be used to evaluate baseline quality of life for each patient prior to and post intervention period. It has been utilized in patients with low back pain and post lumbar surgeries. A higher score on questionnaire indicates better functioning
Change from Baseline Post Surgery (Quality of life Scale) | 3 months
  The Quality of Life Scale consists of only one item, and is utilized to obtain a general quality of life assessment.Scores can range from 16 to 112. Higher scores shows higher quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Professor Amer Aziz, Study Chair — Ghurki Trust and Teaching Hospital
Locations (1):
- Ghurki Trust and Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No